CLINICAL TRIAL: NCT02730065
Title: Effects of Aerobic Dance Training on Cognitive Functions, Mood and Physical Functions in Community Elderly Persons With Cerebral Small Vessel Disease
Brief Title: Aerobic Dance Training in Small Vessel Disease
Acronym: ADTSVD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Adrian Wong, Research Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 03140936
Record Dates: First submitted 2016-03-06; First posted 2016-04-06 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Cerebrovascular Disease
Keywords: Cerebral small vessel disease; Lifestyle modification; Physical activity; Primary prevention; Aerobic dance; Cognition; Depression; Activities of daily living; Cerebral autoregulation
MeSH Terms: conditions — Cerebrovascular Disorders; Cerebral Small Vessel Diseases; Motor Activity; Depression | interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Structured Aerobic Dance Training Group (Active Comparator): Active intervention will last for 24 weeks and consists of 60-minute/session, which includes 10 minutes warm-up, 40 minutes of dancing and 10 minutes of cool down. In groups of 5, participants will practice the dance led by a physiotherapist once per week for the first 2 months and twice per week for 3rd to 6th month.
  Interventions: Behavioral: Structured Aerobic Dance Training Group
- Stretching plus education (Placebo Comparator): Participants in the control group will receive a weekly 3-hour group-based (group of 5 participants) programme containing stretching exercise, stress reduction and health education on dementia and stroke prevention for 6 months. The programme consists of low-intensity seated stretching, psychoeducation on stress management, various relaxation methods with practice as well as education on the causes, identification, treatment and prevention of stroke and dementia. Benefits of physical exercise will also be discussed but will its weight will be evenly balanced with other forms of evidence-based preventive strategies.
  Interventions: Behavioral: Stretching plus education

INTERVENTIONS:
Behavioral: Structured Aerobic Dance Training Group — Systematic physical activity
  Arms: Structured Aerobic Dance Training Group
Behavioral: Stretching plus education — Weekly group based stretching with psychoeducation and health education
  Arms: Stretching plus education

SUMMARY:
Introduction: Cerebral small vessel disease (SVD) is associated with age-related disabilities including dementia, depression, physical and functional impairment. Chinese are more prone to developing SVD than Caucasians. Physical exercise may improve multiple negative consequences associated with SVD.

Objective and hypothesis to be tested: To examine the effects of a 24-week structured aerobic dance training on cognition, mood, physical and daily functions in stroke and dementia free older adults with SVD, and whether such effects are mediated through improved cerebral vasomotor reactivity (CVR), a marker of cerebral autoregulation which is impaired in SVD.

Design and subjects: Rater-blind RCT comparing the effects of 24-week of structured aerobic dance training upon cognition, mood, physical and daily functions on 110 community dwelling, stroke- and dementia-free persons aged ≥65 with MRI evidence of significant SVD, defined as the presence of multiple (≥2) lacunes and/or early confluent or confluent WML.

Interventions: Participants are randomized in a 1:1 ratio into a 24-week of structured therapist-led group aerobic dance training with home practice or simple stretching plus health education control group.

Main outcome measures: Cognition, mood, physical and daily functions and CVR measured using Transcranial Doppler at baseline, weeks 12, 24 and 36.

Data analysis: Intent-to-treat with multiple imputations with treatment efficacy analyzed using mixed effects models. Mediation effects of CVR between aerobic dance training and treatment outcomes tested using mediation models.

Expected results: In persons with significant SVD, aerobic dance training improves cognitive, mood, physical and daily functions and such effects are mediated by changes in CVR.

DETAILED DESCRIPTION:
Cerebral small vessel disease (SVD) is manifested as age-related white matter lesions (WML) and lacunar infarcts and on brain imaging. SVD is prevalent in the elderly population. In community dwelling persons ≥ 60 years of age, up to a quarter had lacunar infarcts and 96% had varying degree of WML. Significant SVD, namely early confluent or confluent WML and multiple lacunar infarcts, are found in up to 1 in every 5 elderly persons. In a previous study we found that Chinese are more prone to develop significant SVD than Caucasians. SVD is associated with a plethora of age-related disabilities such as dementia, falls, depression, impaired daily functioning and death Cognition - SVD is the most common cause of vascular cognitive impairment (VCI) and vascular dementia, which is the second most prevalent type of dementia. Community elderly persons with SVD had two-fold increased risk of developing dementia when compared to those without. SVD may direct damage neural structures, disrupt connectivity or cause atrophy in brain regions important for cognitive functioning. Depression - Disconnection of frontosubcortical pathways by SVD contributes to late-life depression, and increased comorbidity of depression and SVD has been observed in the older populations. Depression contributes to poor quality of life and death in older persons.

Physical impairment - increased severity of SVD is associated with poor physical functions including poor gait and balance. SVD is a strong risk factor for falls, a major contributing factor for disability and death in older persons. In summary, non-disabled older adults with SVD are at high risk of multiple disabilities.

As the elderly population in Hong Kong is projected to triple over the next 30 years, means to prevent age-related disabilities such as cognitive decline, depression and physical impairments in vulnerable individuals are of enormous importance to the patient, family and healthcare system. Existing preventive therapies mainly involve medications to control vascular risk factors associated with SVD. Primary prevention by means of lifestyle intervention is therefore of utmost importance.

Evidence on effects of physical activities upon cognition, mood and physical functions The health values of physical activities are well recognized. Physical activities can be performed by anybody at any time and place at minimal cost. Physical activities are shown to improve the clinical conditions associated with SVD. For cognition, physical activities are associated with reduced risk of cognitive decline in normal and cognitively impaired elderly persons. Aerobic and strength training improved executive functions, memory and general cognitive functions in community-dwelling adults with mild cognitive impairment. The investigators showed that in a large cohort (n=1,013) of stroke patients free of dementia before the stroke, participation in regular physical activities reduced 79% of risk of incident dementia after stroke. With regard to the mechanism, physical activities may improve endothelial functions and blood perfusion and neuroplasticity in brain regions mediating cognitive functions. Moreover, physical exercise may protect cognition by reducing incident strokes, which is particular relevant to people with SVD due to their increased risk of strokes. A randomized controlled trial (RCT) showed that a 24-week, 3 x 50-minute per week of moderate intensity exercise intervention significantly improved cognitive functions in patients at risk of AD, with outcome effect size superior to that reported for drug treatment in another study. Moreover, treatment benefits persisted at least one year after active intervention, suggesting that physical exercise is associated with enduring changes in the neurological substrate underpinning cognitive functioning. However, this study only recruited patients likely to have degenerative (Alzheimer's) pathology. For mood, physical activities may protect against depression in older adults. For physical functions, the investigators previously showed that physical exercise training improved balance, gait performance, exercise endurance and quality of life in local patients with Parkinson's Disease (PD). Taken together, there is good evidence that physical activities can improve many of the negative consequences of cerebral SVD.

Possible biological mechanism underlying physical exercise in SVD The development of SVD is hypothesized to be related to endothelial dysfunction that results from chronic hypertension impairs cerebral vasomotor reactivity (CVR), a marker of cerebral autoregulation. Changes in CVR may reflect impairment in the homeostasis of blood pressure in the brain, hence cerebral perfusion becomes more dependent on the systemic blood pressure. Ischemia occurs in response to drop of systemic blood pressure and lead to hypoperfusion and subsequently the development of SVD. Using Transcranial Doppler (TCD) ultrasonography, our group previously showed that decreased CVR is associated with SVD. Reduced CVR is linked to cognitive decline, depression and poor physical functions in elderly persons. Physical exercise may lead to significant improvement in CVR. These data suggest that physical exercise is likely to benefit cognition, mood and physical functions in persons with SVD due to its positive effects on CVR.

Dancing as a mean of physical activity intervention Dance is a rhythmic movement usually performed with music. To many, it is a pleasurable activity that can be taken up as a hobby and social activity and therefore engagement can be self-sustaining. It is of minimal-cost and can be performed even in older persons with physical and cognitive impairment. Dancing involves movement of the body and limbs and is in itself a physical training. It also involves memory, attention, sensory stimulation, social interaction, emotional perception and expression that presumably could protect against cognitive decline and depression. Dance training may improve verbal fluency, word list delayed recall and word list recognition in older adults with metabolic syndrome, suggesting that dance may be effective in preventing cognitive decline. Aerobic dance also has been shown to enhance exercise endurance strength, balance, agility and gait performance in older adults. Our team had previously designed and implemented a balance dance to a group of patients with PD for 8 weeks. Together with other training, balance ability and walking speed increased and the effects lasted for 12 months after treatment completion. Given the likely positive effects of aerobic dance, it appears to be a good exercise candidate for enhancing cognitive, mood and physical functions in patients with cerebral SVD.

Data Collection Assessment of cognitive functions The 30-minute protocol of the National Institute of Neurological Diseases and Stroke - Canadian Stroke Network VCI protocols will be used. The 30-minute protocol provides a comprehensive assessment of cognitive functions with emphasis on executive functions, psychomotor speed and memory, which are the cognitive domains predominately impaired in VCI. With support from Health and Health Service Research fund (PI: Vincent CT MOK; Reference Number 06070231), the investigators adapted and validated the 30-minute protocol in a group of Chinese stroke patients and controls and demonstrated good external validity (area under ROC=0.79 [95%CI 0.69-0.89], p<0.001) in differentiating stroke patients from non-stroke controls and concurrent validity with functional measures. In addition to the 30-minute protocol, the digit span tests from the Wechsler Memory Scale will be administered because of the involvement of immediate attention and working memory in VCI.

Measure of depressive symptoms The 15-item Geriatric Depression Scale (GDS), which is a self-reported questionnaire to rate depressive symptoms in elderly persons, will be used. It has been used in local study on SVD patients and demonstrated excellent classification power >90% in detecting depression in the local elderly population.

Measures of physical functions The Mini-Balance Evaluation Systems Test (Mini-BESTest) will be used to assess dynamic balance performance of individuals. The 14-item Mini-BESTest represents 4 dynamic balance domains: anticipatory postural adjustments, postural responses, sensory orientation and stability in gait. Each item is rated from 0 to 2, and the total score ranges from 0-28 with a higher score indicating better balance.

The Timed-up-and-go test (TUG) will be used to examine functional mobility of subjects. This test measures the time which participants takes to rise from the chair, walk 3 meters, turn around, walk back to the chair and sit down.

The 6-minute walk test will be used to determine the walking capacity. This test measures the distance (in metres) participants walk in 6 minutes. Participants will walk at their own speed, and stops and resting are allowed if necessary.

Measure of daily functions The Lawton's Instrumental Activities of Daily Living (IADL) will be used to assess complex activities of daily functions that are impaired early in patients with SVD. It take about 10 minutes to administer and contains 8 items including ability to use telephone, shopping, food preparation, housekeeping, laundry, taking transportation, handling medications and finances. It is has been used as a primary outcome instrument in the Pan-European Leukoaraiosis and Disability in the Elderly Study in SVD.

Measure of overall physical activities Physical activities performed outside of training session will be recorded using the long form of the International Physical Activity Questionnaire (IPAQ). The IPAQ has been very widely used in studies of physical activity across different ages and medical conditions (http://www.ipaq.ki.se/publications.htm). The IPAQ records the types, frequency and duration of physical activities across 4 activity domains including leisure time physical activity, domestic related physical activities, work-related and transportation related physical activities. The IPAQ yields scores for walking, moderate-intensity and vigorous-intensity activities with each of these activity domains. A total score is calculated by summing the duration and frequency for all types of activities across all domains. This score will be used to account for the potential confounding effects of physical activities performed outside of training session in both groups.

It is estimated that it takes approximately 2 hours to complete the assessment and TCD examination. To avoid rater bias, the research assistant (RA) who performs the study assessment will be blind to treatment allocation and encouraged not to discuss with the participants about the interventions. Clinical assessments will be performed by a trained RA under the supervision of a qualified clinical psychologist (PI of this application).

TCD Examination TCD examination will be performed at baseline, weeks 12, 24 and 36. A 2-MHz pulsed Doppler hand-held probe is used to insonate the middle cerebral artery (MCA) through temporal window above the zygomatic arch at a depth of 52-56mm, and the vertebral artery (VA) through occipital window at a depth of 64mm. The Pulsatility Index (PI) and Breath Holding Index (BHI) will be calculated. The PI is a measure of vascular resistance of cerebral vessels. The mean PI of the middle MCA and vertebral VA will be obtained. A previous study by the investigators showed that these measures highly differentiated stroke patients with and without WML on MRI (AUC = 0.85 [MCA] and 0.81 [VA], sensitivity and specificity between 70 and 82%]). According to the standard protocol, the simple breath holding procedure will be performed during the same TCD session to obtain the BHI, which will serve as a marker of CVR. A trained postgraduate research student under the supervision of a broad certified neurologist (Co-A Vincent MOK) will perform the TCD blind to participant's treatment allocation.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥65
2. Community dwelling
3. Presence of significant SVD, defined by the presence of multiple (≥2) lacunar infarcts and/or a rating of ≥2 (i.e. beginning confluence of lesions to diffuse involvement of lesions in periventricular and/or deep white matter) of WML using the Age-related White Matter Changes (ARWMC) Scale on MRI
4. Presence of good temporal window on at least one side for TCD evaluation
5. Written informed consent given

Exclusion Criteria:

1. History of stroke
2. Dementia, determined by a score on Cantonese MMSE less than education adjusted cutoff score for dementia or history of dementia diagnosis
3. Comorbidity with medical conditions affecting the central nervous system or cerebral white matter
4. Inadequately controlled psychiatric disorders affecting cognition and mood
5. Physical or sensory impediments hindering participation in cognitive assessment or exercise training.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Cognition assessed by the 30-minute protocol of the National Institute of Neurological Diseases and Stroke - Canadian Stroke Network VCI protocol summary score | Change from baseline to week 24
Depressive symptoms evaluated the Geriatric Depression Scale | Change from baseline to week 24
Physical balance measured by the Mini-Balance Evaluation Systems Test | Change from baseline to week 24
Functional mobility measured by the Timed-up-and-go test | Change from baseline to week 24
Walking capacity assessed by the 6-minute walk test | Change from baseline to week 24
Daily functioning evaluated by the Lawton's Instrumental Activities of Daily Living | Change from baseline to week 24

SECONDARY OUTCOMES:
Cerebral vasomotor reactivity measured by Pulsatility Index obtained from middle cerebral artery and vertebral artery measured on Transcranial Doppler | Change from baseline to week 24
Cerebral vasomotor reactivity measured by Breath Holding Index obtained from middle cerebral artery and vertebral artery measured on Transcranial Doppler | Change from baseline to week 24

OTHER OUTCOMES:
Number of participants with adverse events or serious adverse events | Throughout the entire study period up to 36 weeks
  Adverse events and serious adverse events will be reported to the Chinese University of Hong Kong - New Territories East Cluster Ethics Committee according to standard reporting guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Wong, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Chinese University of Hong Kong, Hong Kong
  - Neurology Clinical Research Centre, CUHK, Shatin

IPD SHARING:
Plan to Share IPD: Undecided